CLINICAL TRIAL: NCT05698771
Title: NAD-brain: a Pharmacokinetic Study of NAD Replenishment Therapy
Acronym: NAD-brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-496197
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: nicotinamide adenine dinucleotide; NAD; NAD+; pharmacokinetics; nicotinamide riboside; nicotinamide mononucleotide; brain kinetics
MeSH Terms: interventions — nicotinamide-beta-riboside; Nicotinamide Mononucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NR Stage-1 Healthy (Experimental): A total of 6 individuals comprising 3 males and 3 females will receive NR 1200 mg daily (600 mg x 2) for 8 days, with a total measurement/assessment period of 20 days. These will be the same individuals as in the NMN-arm. The individuals will enter the two arms sequentially and with a washout period of 14 days.
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- NMN Stage-1 Healthy (Experimental): A total of 6 individuals comprising 3 males and 3 females will receive NMN 1200 mg daily (600 mg x 2) for 8 days, with a total measurement/assessment period of 20 days. These will be the same individuals as in the NR-arm. The individuals will enter the two arms sequentially and with a washout period of 14 days.
  Interventions: Dietary Supplement: nicotinamide mononucleotide
- NR Stage 2 Healthy (Experimental): A total of 6 healthy individuals (3 men and 3 women) will receive NR 1200 mg daily (600 mg x 2) for for 4 weeks, followed by 3 weeks of washout (total period of follow-up is 7 weeks).
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- NR Stage-2 Parkinson's disease (Experimental): A total of 6 with Parkinson's disease (3 men and 3 women) will receive NR 1200 mg daily (600 mg x 2) for for 4 weeks, followed by 3 weeks of washout (total period of follow-up is 7 weeks).
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — The NAD-brain study will perform a parallel assessment of NAD replenishment therapy (NRT) pharmacokinetics in the blood and brain of healthy human subjects . A total of 6 healthy individuals (3 men and 3 women) will undergo repeated blood sampling and 31P-MRS brain scans during two 20-day periods, each of which will start with 8 days of daily intake of Nicotinamide Riboside (NR) 600mg x 2, or Nicotinamide Mononucleotide (NMN) 600mg x 2. The two 20-day periods will be 14 days apart to allow for washout of the previous compound. Blood will be analyzed for NAD-metabolites using spectroscopic assays. By this approach we will measure the simultaneous change in NAD-metabolism over time in blood and brain and establish blood and brain pharmacokinetics for NRT in humans.
  Other Names: NR Stage-1 Healthy
  Arms: NR Stage-1 Healthy
Dietary Supplement: nicotinamide mononucleotide — The NAD-brain study will perform a parallel assessment of NAD replenishment therapy (NRT) pharmacokinetics in the blood and brain of healthy human subjects. A total of 6 healthy individuals (3 men and 3 women) will undergo repeated blood sampling and 31P-MRS brain scans during two 20-day periods, each of which will start with 8 days of daily intake of Nicotinamide Riboside (NR) 600mg x 2, or Nicotinamide Mononucleotide (NMN) 600mg x 2. The two 20-day periods will be 14 days apart to allow for washout of the previous compound. Blood will be analyzed for NAD-metabolites using spectroscopic assays. By this approach we will measure the simultaneous change in NAD-metabolism over time in blood and brain and establish blood and brain pharmacokinetics for NRT in humans.
  Other Names: NMN Stage-1 Healthy
  Arms: NMN Stage-1 Healthy
Dietary Supplement: Nicotinamide Riboside (NR) — A total of n=6 healthy individuals (3 men and 3 women) will receive NR 1200 mg per day for 4 weeks, followed by 3 weeks of washout. The individuals will undergo repeated blood sampling and 31P-MRS brain scans once per week during the 7 weeks period, Blood will be analyzed for NAD-metabolites using spectroscopic assays.
  Other Names: NR Stage-2 Healthy
  Arms: NR Stage 2 Healthy
Dietary Supplement: Nicotinamide Riboside (NR) — A total of n=6 individuals with Parkinson's disease (3 men and 3 women) will receive NR 1200 mg per day for 4 weeks, followed by 3 weeks of washout. The individuals will undergo repeated blood sampling and 31P-MRS brain scans once per week during the 7 weeks period, Blood will be analyzed for NAD-metabolites using spectroscopic assays.
  Other Names: NR Stage-2, Parkinson's disease
  Arms: NR Stage-2 Parkinson's disease

SUMMARY:
The objective of the NAD-brain study is to determine the blood and brain pharmacokinetics of NAD replenishment therapy (NRT) using Nicotinamide Riboside (NR) or Nicotinamide Mononucleotide (NMN).

DETAILED DESCRIPTION:
The NAD-brain study will perform a parallel assessment of NAD replenishment therapy (NRT) pharmacokinetics in the blood and brain of healthy human subjects. A total of 6 healthy individuals (3 men and 3 women) will undergo repeated blood sampling and 31P-MRS brain scans during two 20-day periods, each of which will start with 8 days of daily intake of Nicotinamide Riboside (NR) 600mg x 2, or Nicotinamide Mononucleotide (NMN) 600mg x 2. The two 20-day periods will be 14 days apart to allow for washout of the previous compound.

Moreover, a total of 6 healthy individuals (3 men and 3 women) and 6 individuals with Parkinson's disease (3 men and 3 women) will receive NR 1200 mg daily (600 mg x 2) for 4 weeks, with a total measurement/assessment period of 7 weeks, and undergo repeated blood sampling and 31P-MRS brain scans once per week during this time.

Blood will be analyzed for NAD-metabolites. The simultaneous change in NAD-metabolism over time in blood and brain will be assessed and blood and brain pharmacokinetics for NRT in humans will be established.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-85 years at the time of enrollment.
* Neurologically healthy at the time of enrollment.

Exclusion Criteria:

* History of acute or chronic neurological disorder affecting the central nervous system (CNS). Migraine, cluster headache, and tension headache are allowed, but not on the day of the study visits.
* Impaired renal function.
* Impaired hepatic function.
* Severe hematological disease.
* Any psychiatric disorder that would interfere with compliance in the study.
* Any severe somatic illness that would make the individual unable to comply and participate in the study.
* Mitochondrial disease.
* Use of high dose vitamin B3 supplementation within 30 days of enrolment.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
NAD metabolism | For Stage-1: 20 days for NR and 20 days for NMN comprising 8 days treatment, and 11 days washout. For Stage-2 (NR): 7 weeks comprising 4 weeks of treatment and 3 weeks washout
  The change of cerebral NAD levels (measured by 31P-MRS) and of blood NAD-metabolites (measured by HPLC-MS), over time (20 days), after the administration of oral NRT with the following NAD precursors: NR 600mg x 2 daily, NMN 600mg x 2 daily.

SECONDARY OUTCOMES:
Interindividual differences | For Stage-1: 20 days for NR and 20 days for NMN comprising 8 days treatment, and 11 days washout. For Stage-2 (NR): 7 weeks comprising 4 weeks of treatment and 3 weeks washout
  Descriptive analyses of interindividual differences in the time course of change in the blood NAD-metabolome and cerebral NAD increase, following the administration of oral NRT.
Between-sex differences | For Stage-1: 20 days for NR and 20 days for NMN comprising 8 days treatment, and 11 days washout. For Stage-2 (NR): 7 weeks comprising 4 weeks of treatment and 3 weeks washout
  Between-sex differences in the time course of change in the blood NAD-metabolome and cerebral NAD increase, following the administration of oral NRT.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, MD, PhD, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No